CLINICAL TRIAL: NCT01364610
Title: A Prospective Assessment of pH Testing Methods in Alberta
Brief Title: An Assessment of pH Testing Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Christopher Andrews, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Bravo
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Gastroesophageal Reflux
Keywords: diagnosis; pH measurement; catheter; wireless
MeSH Terms: conditions — Gastroesophageal Reflux; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Active Comparator): Group 1 will have standard catheter based pH-metry. All participants will answer a questionnaire assessing tolerance and satisfaction of both the siting and placement methods and the 24 hour monitoring period.
  Interventions: Device: Standard Care
- Bravo pH Monitoring System (Active Comparator): Group 2 will undergo unsedated peroral placement of the Bravo capsule. All participants will answer a questionnaire assessing tolerance and satisfaction of both the siting and placement methods and the 24 hour pH monitoring period.
  Interventions: Device: Bravo

INTERVENTIONS:
Device: Bravo — Bravo pH Monitoring System sited manometrically.
  Other Names: Bravo pH Monitoring System
  Arms: Bravo pH Monitoring System
Device: Standard Care — Nasally passed pH catheter sited by manometry, accompanied by battery powered data logger. Participant activated event marker in response to symptoms, meals and body position changes.
  Arms: Standard Care

SUMMARY:
Gastroesophageal reflux disease (GERD) is a common and potentially debilitating disorder. Typical symptoms include heartburn and regurgitation of acid tasting substances. GERD is a chronic disease and in some cases, more alarming symptoms including food sticking in the esophagus, pain with swallowing, bleeding, anemia and weight loss develop.

In Alberta, upper endoscopy is the first line of investigation accompanied by an ambulatory 24-hour esophageal pH monitoring for patients with symptoms that are unresponsive to acid-suppressing therapy or who exhibit alarm symptoms.

Current standard of care in Alberta for esophageal pH monitoring first requires an esophageal manometry test to identify the location of the lower esophageal sphincter followed by the placement of a thin catheter with one or more pH probes inserted through the nose and taped in place to the face for 20 -24 hours. The patient wears a small battery powered data logger and maintains a diary of GERD symptoms and activity. This system enables the recording and correlation of specific symptoms with reflux episodes over extended periods and provides direct evidence of GERD. The nasally passed pH catheter is uncomfortable and restrictive for some patients often resulting in abnormal eating, drinking, activity and sleeping patterns. The data collected may not be representative of the patient's typical experience and may not reflect the true severity of the disease.

A wireless diagnostic pH monitoring system called Bravo pH Monitoring System developed by Medtronic is approved for use in Canada and is commercially available. This system eliminates the need for a catheter by utilizing a capsule the size of a gel-cap and radio frequency technology to monitor esophageal pH. It has been shown to be safe and as sensitive as conventional catheter-based pH probe monitoring. The Bravo system can be sited either endoscopically or manometrically.

The goal of this study is to test the Bravo Wireless pH system in Alberta using manometric siting to assess feasibility, patient outcomes and tolerance.

Hypotheses:

1. Patient tolerance of the Bravo system is superior to standard pH-metry.
2. Manometric placement of Bravo is as successful as standard pH-metry.

Our aims:

1. To assess patient tolerance of Bravo versus standard pH-metry.
2. To compare the success rate of manometric peroral placement of Bravo pH probe versus standard pH-metry.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years
* Able to provide written consent
* Symptoms potentially due to acid reflux and referred for an ambulatory pH study as part of routine clinical care
* Able and willing to potentially undergo peroral Bravo placement
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study

Exclusion Criteria:

* Previous esophageal surgery, or any known anatomic or functional defect of the digestive tract that might make capsule passage or retrieval unsafe
* Clinical evidence (including physical exam and/or EKG) of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric or other disease that may interfere with the objectives of the study and/or pose safety concerns
* Allergy to topical anesthetic
* Any implanted electrical device such as a pacemaker, defibrillator or neurostimulator
* Pregnant or breast-feeding females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Overall discomfort with standard vs. Bravo pH-metry. | 24 hours
  Mean overall discomfort from the pH-metry procedure between Group 1 (standard) and Group 2 (Bravo) as measured by questionnaire.

SECONDARY OUTCOMES:
Success rate of Bravo capsule placement | 24 hours
  As defined by completion of the manometry to find the Bravo placement depth; completion of peroral Bravo placement; adequate deployment and adherence of the Bravo capsule to the esophageal mucosa for a minimum of 20 hours.
Site specific discomfort of both siting and placement procedures | 24 hours
Ability to do normal activities | 24 hours
Time off work | 24 hours
  Difference in recorded time off work for Group 1 (standard) vs. Group 2 (Bravo)
Procedure Related Costs | 24 hours
  Procedure related costs between groups (including primary payer and societal costs)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

REFERENCES:
- [Derived] Andrews CN, Sadowski DC, Lazarescu A, Williams C, Neshev E, Storr M, Au F, Heitman SJ. Unsedated peroral wireless pH capsule placement vs. standard pH testing: a randomized study and cost analysis. BMC Gastroenterol. 2012 May 31;12:58. doi: 10.1186/1471-230X-12-58. PMID 22650250